CLINICAL TRIAL: NCT02391961
Title: Study and Treatment of Visual Dysfunction and Motor Fatigue in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: F1180-W; 1IK2RX001180-01A2 (NIH)
Record Dates: First submitted 2015-03-03; First posted 2015-03-18 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Multiple Sclerosis; Internuclear Ophthalmoplegia; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Ocular Motility Disorders; Fatigue | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dalfampridine (Experimental): 10-week randomized, placebo controlled, double-blind, crossover trial, which includes a period of wash out of two weeks between treatment with dalfampridine and placebo. Within the trial, each patient serves as his own control.
  Interventions: Drug: Dalfampridine
- placebo (Placebo Comparator): 10-week randomized, placebo controlled, double-blind, crossover trial, which includes a period of wash out of two weeks between treatment with dalfampridine and placebo. Within the trial, each patient serves as his own control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dalfampridine — 10-week randomized, placebo controlled, double-blind, crossover trial, which includes a period of wash out of two weeks between treatment with dalfampridine and placebo.
  Arms: dalfampridine
Drug: Placebo — 10-week randomized, placebo controlled, double-blind, crossover trial, which includes a period of wash out of two weeks between treatment with dalfampridine and placebo.
  Arms: placebo

SUMMARY:
Primary fatigue represents a major cause of disability in patients with multiple sclerosis (MS), being reported in about 90% of cases. Fatigue interferes with everyday functioning but, unfortunately, little is known about its mechanisms. The investigators propose a characteristic eye movement abnormality (internuclear ophthalmoparesis, INO), commonly encountered in MS, as a simple model for primary motor fatigue. The investigators described worsening of ocular performance in MS patients with INO following visual tasks (ocular motor fatigue), which is likely due to decreased neural conduction along brain pathways injured by MS. This mechanism could represent a major component of MS-related primary motor fatigue. Relevant to Veterans' care, INO is a significant cause of visual disability, especially when complicated by ocular fatigue, and limits daily activities such as reading and driving. The investigators propose a medical treatment to improve ocular performance/fatigue in INO, which can reduce visual disability and improve quality of life in Veterans with MS.

DETAILED DESCRIPTION:
This project focuses on fatigue, an extremely common yet poorly understood complaint in patients affected by multiple sclerosis (MS). Primary fatigue, that is fatigue not secondary to other MS-associated symptoms (e.g., sleep disorder or depression), is a distinct clinical entity and a cause of severe disability in most patients. As fatigue limits everyday activities and interferes with exercise-based rehabilitation, understanding its mechanisms is crucial to improving function and quality of life of Veterans with MS. Primary fatigue is divided in two broad categories, mental (cognitive) and physical (motor) fatigue, the latter being the focus of this proposal. Evidence suggests that primary motor fatigue originates within the central nervous system (CNS) but, although several factors have been invoked (e.g., demyelination, axonal loss, inflammation), a neurophysiological model to explain its underlying mechanisms is still lacking.

First, with this project, the investigators propose a characteristic eye movement abnormality, internuclear ophthalmoparesis (INO), as a simple and accessible model for primary motor fatigue in MS. INO is a disorder of binocular coordination (conjugacy), in which fast eye movements (saccades) of the adducting eye (i.e., the eye moving towards the nose) are slow during horizontal gaze shifts, due to demyelination of a specific CNS pathway (the medial longitudinal fasciculus, MLF). Preliminary results in a small MS group of patients show that patients with INO exhibit changes in ocular conjugacy (i.e., ocular motor fatigue) during a 10-minute saccadic fatigue test, but normal subjects do not. The investigators hypothesize that ocular motor fatigue is representative of a major component of primary motor fatigue in MS, as it likely reflects deterioration of neural conduction fidelity along the demyelinated MLF axons. The investigators aim at showing that ocular motor fatigue occurs in a larger MS population with INO by measuring changes of binocular conjugacy on eye movement recordings using two main measures: 1) abducting/adducting eye ratio for saccadic peak velocity (pulse size ratio); 2) time difference in occurrence of peak acceleration in the adducting vs. the abducting eye (pulse time delay), during the 10-minute fatigue test. The investigators will determine whether ocular motor fatigue is associated with symptomatic subjective fatigue as assessed with standard fatigue questionnaires. Second, The investigators intend to test efficacy of dalfampridine, a potassium channel blocker that enhances neural conduction along demyelinated axons, in MS patients with INO with or without associated ocular motor fatigue. Visual dysfunction in MS patients with INO is a major cause of disability as they are severely limited in daily activities such as driving and can suffer further disability when developing ocular motor fatigue during a sustained visual task (e.g., reading). However, no medical therapy is available for INO/ocular motor fatigue. Preliminary results document improved binocular conjugacy in three MS patients taking dalfampridine for gait impairment (the FDA-approved indication for this medication). These data also showed improvement of ocular motor fatigue after dalfampridine in one patient. The investigators hypothesize that dalfampridine improves visual performance in MS patients with INO and counteracts ocular motor fatigue and, in turn, diminishes visual disability and improves quality of life. Thus, the investigators will conduct a randomized, placebo-controlled, double-blind, crossover trial of dalfampridine (10mg twice a day) of 10 weeks duration. Before and after treatment, the investigators will assess for changes in binocular conjugacy by eye movement measures as above, as well as changes in clinical measures, such as reading acuity and speed, saccades performance, gait performance, symptomatic fatigue, visual disability and quality of life. the investigators will determine whether improvement of visual performance has positive effects on overall disability and quality of life of MS patients with INO. The investigators will also determine whether there is an association between response of eye movement and gait performances to dalfampridine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS of any course and duration
* Evidence of mild to moderate internuclear ophthalmoparesis (INO), that is slowing of the adducting eye on physical examination of saccadic speed, whether INO is unilateral or bilateral, symmetrical or asymmetrical
* Medically stable conditions, ability to give informed consent and understand and cooperate with the testing
* Dalfampridine-naive as well as history of taking dalfampridine in the past, whether there was benefit in gait impairment or not, after a washout period of at least 2 weeks

Exclusion Criteria:

* Lack of evidence of INO (slowing of the adducting eye) on physical examination of saccadic speed
* Severe INO (i.e., exotropia in primary gaze) on physical examination
* Medically unstable conditions, inability to give informed consent and understand and cooperate with the testing
* History of side effects from dalfampridine
* History of seizures
* Moderate or severe renal failure, assessed by clearance of creatinine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Serra, MD PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra A, Chisari CG, Matta M. Eye Movement Abnormalities in Multiple Sclerosis: Pathogenesis, Modeling, and Treatment. Front Neurol. 2018 Feb 5;9:31. doi: 10.3389/fneur.2018.00031. eCollection 2018. PMID 29467711

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: (4) subjects were enrolled, but did not pass initial screening procedures at study visit 1 and therefore were not assigned to a study group.
Groups:
- Dalfampridine, Then Placebo: Participants were randomized to receive dalfampridine 10 mg tablet twice a day for 4 weeks (First Intervention) then, after a washout period of 2 weeks, did receive placebo tablet twice a day (matching dalfampridine 10 mg tablet) for 4 weeks (Second Intervention).
- Placebo, Then Dalfampridine: Participants were randomized to receive placebo tablet (matching dalfampridine 10 mg tablet) twice a day for 4 weeks (First Intervention) then, after a washout period of 2 weeks, did receive dalfampridine 10 mg tablet twice a day for 4 weeks (Second Intervention).
Period: First Intervention (4 Weeks)
Arm/Group | Dalfampridine, Then Placebo | Placebo, Then Dalfampridine
Started | 10 | 9
Completed | 8 | 9
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Washout (2 Weeks)
Arm/Group | Dalfampridine, Then Placebo | Placebo, Then Dalfampridine
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention (4 Weeks)
Arm/Group | Dalfampridine, Then Placebo | Placebo, Then Dalfampridine
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Because Internuclear Ophthalmoparesis (INO) was bilateral in some participants, the overall number of INO was different than the number of participants.
Units Other Than Participants: INO
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalfampridine, Then Placebo | Placebo, Then Dalfampridine | Total
Number analyzed (Participants) | 10 | 9 | 19
Number analyzed (INO) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (8.5) | 47.8 (11.2) | 47.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pulse Size Ratio (PSR): Abducting/Adducting Eye Ratio for Saccadic Peak Velocity.
Description: For each saccade made by the subject, the ratio of the maximum velocity (deg/sec) of the eye moving away from the nose and of the eye moving towards the nose was calculated. Subjects' horizontal saccades were recorded for 10 minutes, and an average of PSR for all saccades recorded was taken.
Time Frame: Average PSR values were taken on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks), on each visit before (baseline) and three hours after taking the study pill.
Population: Some participants withdrew after visit 1, visit 2 or 3. (1) more participant was not included in the final analysis as missing a datapoint (baseline data at Visit 2). Thus, the number above (12) is the number of participants who completed the full protocol from visit 1 to visit 4.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: INO (internuclear ophthalmoparesis)
Groups:
- Dalfampridine: Participants were randomized to receive dalfampridine 10 mg or placebo tablet twice a day for 4 weeks (First Intervention) then, after a washout period of 2 weeks, did receive dalfampridine 10 mg or placebo tablet twice a day for 4 weeks (Second Intervention), according to the trial crossover design.
  Here we report results from participants while on dalfampridine.
- Placebo: Participants were randomized to receive dalfampridine 10 mg or placebo tablet twice a day for 4 weeks (First Intervention) then, after a washout period of 2 weeks, did receive dalfampridine 10 mg or placebo tablet twice a day for 4 weeks (Second Intervention), according to the trial crossover design.
  Here we report results from participants while on placebo.
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
Number analyzed (INO (internuclear ophthalmoparesis)) | 20 | 20
ratio
  average pulse size ratio baseline | 1.914 (0.454) | 1.937 (0.553)
  average pulse size ratio after 3 hours | 1.805 (0.451) | 1.898 (0.508)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 4 subgroups: average PSR at baseline and after 3 hours on dalfampridine, and average PSR at baseline and after 3 hours on placebo; Test type: Superiority; p = 0.842672, ANOVA

2. Primary Outcome: Pulse Time Delay (PTD): Time Difference Between Onset of the Saccade in the Adducting Eye and Onset of the Saccade in the Abducting Eye.
Description: For each saccade made by the subject, we calculated the difference (in sec) between the onset (based on a velocity threshold) of the movement in the adducting eye (the eye moving towards the nose) and the onset of the movement in the abducting eye (the eye moving away from the nose). Subjects' horizontal saccades were recorded for 10 minutes, and an average of PTD for all saccades recorded was taken.
Time Frame: Average PTD values were taken on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks), on each visit before (baseline) and three hours after taking the study pill.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: INO (internuclear ophthalmoparesis)
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
Number analyzed (INO (internuclear ophthalmoparesis)) | 20 | 20
seconds
  Average PTD at baseline | 0.007 (0.005) | 0.007 (0.005)
  Average PTD after 3 hours | 0.008 (0.004) | 0.008 (0.004)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 4 subgroups: average PTD at baseline and after 3 hours on dalfampridine, and average PTD at baseline and after 3 hours on placebo; Test type: Superiority; p = 0.972866, ANOVA

3. Secondary Outcome: Reading Acuity (RA)
Description: MNREAD acuity charts for reading acuity (RA)
Time Frame: Average RA values were taken on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks), on each visit before (baseline) and three hours after taking the study pill.
Measure: Mean (Standard Deviation); unit: logMAR for RA
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
logMAR for RA
  RA at baseline | 0.111 (0.117) | 0.108 (0.138)
  RA after 3 hours | 0.088 (0.121) | 0.086 (0.141)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 4 subgroups: RA at baseline and after 3 hours on dalfampridine, and RA at baseline and after 3 hours on placebo; Test type: Superiority; p = 0.95, ANOVA

4. Secondary Outcome: Maximum Reading Speed (MRS)
Description: MNREAD acuity charts for reading speed (maximum reading speed, MRS)
Time Frame: Average MRS values were taken on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks), on each visit before (baseline) and three hours after taking the study pill.
Measure: Mean (Standard Deviation); unit: words per minute
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
words per minute
  MRS at baseline | 156 (31) | 151.7 (20)
  MRS after 3 hours | 158 (19) | 158.7 (25)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 4 subgroups: MRS at baseline and after 3 hours on dalfampridine, and MRS at baseline and after 3 hours on placebo; Test type: Superiority; p = 0.9, ANOVA

5. Secondary Outcome: Gait Assessment
Description: 25-foot Walk Test (FWT)
Time Frame: Measures were taken on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks), on each visit before (baseline) and three hours after taking the study pill.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
seconds
  25 FWT baseline | 8.986 (4.957) | 9.113 (4.639)
  25 FWT after 3 hours | 8.567 (5.352) | 9.184 (5.400)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 4 subgroups: 25 FWT at baseline and after 3 hours on dalfampridine, and 25 FWT at baseline and after 3 hours on placebo; Test type: Superiority; p = 0.990995, ANOVA

6. Secondary Outcome: National Eye Institute (NEI) Visual Function Questionnaire 25 (VFQ-25)
Description: We used a validated questionnaire to assess visual disability, the National Eye Institute (NEI) Visual Function Questionnaire 25. Min value 0; Max value 100; Higher scores mean a better outcome.
Time Frame: VFQ25 was administered on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | 73.48 (16.65) | 71.62 (22.3)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 2 groups, mean VFQ-25 scores on dalfampridine vs mean VFQ-25 scores on placebo; Test type: Superiority; p = 0.71, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: 10-Item Neuro-Ophthalmic Supplement (NOS)
Description: We used a validated questionnaire to assess visual disability, the 10-Item Neuro-Ophthalmic Supplement. Min value 0; Max value 100; Higher scores mean a better outcome.
Time Frame: 10-Item NOS was administered on day of visit 2 (after 4 weeks) and on day of visit 4 (after 10 weeks).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dalfampridine | Placebo
Number analyzed (Participants) | 12 | 12
score on a scale | 64.9 (24) | 64.3 (25)
Statistical Analysis 1: Comparison: Dalfampridine vs Placebo; Statistical Analysis applies to the 2 groups, mean 10-item NOS scores on dalfampridine vs mean 10-item NOS scores on placebo; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject during their participation time in the study from time of enrollment to study completion or withdrawal, an average of 10 weeks.
Groups:
- Dalfampridine: Participants received dalfampridine 10 mg tablet twice a day for 4 weeks.
- Placebo: Participants received placebo tablet (matching dalfampridine 10 mg tablet) twice a day for 4 weeks.
Arm/Group | Dalfampridine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 2/17 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalfampridine (N=17) | Placebo (N=15)
known mild side effect of medication (Gastrointestinal disorders) | 1 (1) | 0 (0) — the subject reported gastro-intestinal upset with medication use
known side effect of medication (Nervous system disorders) | 1 (1) | 0 (0) — the subject reported insomnia with medication use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02391961/Prot_SAP_000.pdf